CLINICAL TRIAL: NCT06484998
Title: Evaluation Of The Relationship Between Dental Anxiety Levels Of Children And Their Compomer Restoration Colour Preferences
Brief Title: Relationship Between Children's Colour Preferences and Their Dental Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Melek Belevcikli, Assistant professor, Bulent Ecevit University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bülent Ecevit University
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Dental Anxiety; Child Development
Keywords: Colour; Compomer; Dental Anxiety; Dental Caries; Primary teeth
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low anxiety (Experimental): A score was obtained from the MCDASf scale by summing the scores of each question expressed with faces ranging from 1 "relaxed", 2 "slightly worried", 3 "worried", 4 "very worried" and 5 "extremely worried" according to the 8 questions. Those with a total score of less than 19 points were included in this group.
  Interventions: Behavioral: Dental anxiety level and child's compomer colors selection
- moderate anxiety (Experimental): A score was obtained from the MCDASf scale by summing the scores of each question expressed with faces ranging from 1 "relaxed", 2 "slightly worried", 3 "worried", 4 "very worried" and 5 "extremely worried" according to the 8 questions. Those with a total score between 19-31 points were included in this group.
  Interventions: Behavioral: Dental anxiety level and child's compomer colors selection
- high anxiety (Experimental): A score was obtained from the MCDASf scale by summing the scores of each question expressed with faces ranging from 1 "relaxed", 2 "slightly worried", 3 "worried", 4 "very worried" and 5 "extremely worried" according to the 8 questions. Those with a total score between 32-40 points were included in this group.
  Interventions: Behavioral: Dental anxiety level and child's compomer colors selection

INTERVENTIONS:
Behavioral: Dental anxiety level and child's compomer colors selection — Patients without any syndromes or systemic disorders, without mental retardation, who needed restorative treatment for primary molars were included in the study. The examination forms of 275 patients requiring restorative treatment of primary teeth were analysed at the session they came for restorative treatment. To determine the child's anxiety, the Modified Child Dental Anxiety Scale-faces version was administered to the children before restorative treatment. The children were asked to choose from a scale consisting of 9 colours (pink, blue, gold, silver, orange, yellow, green, purple, white) for the compomer restoration color selections. The patients were asked what their favourite color was after the compomer restoration color selection so that the previous question would not have any effect on the child's restoration color selection.

SUMMARY:
The objective of this study was to examine the relationship between children's color preferences and their dental anxiety. It aims to answer are:

1. Is there a relationship between children's compomer restoration colour preferences and dental anxiety?
2. Do children's compomer restoration colour preferences vary according to age and gender?
3. Are children's compomer restoration colour preferences the same as their favourite colours?

DETAILED DESCRIPTION:
Background: Dental fear and anxiety, which are frequently encountered in children, are recognised as an important public health problem in many countries and this situation leads to postponement and neglect of dental treatments. The aim of this study is to evaluate the relationship between colored compomer color preferences and dental anxiety levels, which are frequently used in the restorative treatments of pediatric patients who need restorative treatment of primary molar teeth.

Methods: In this study, the relationship between anxiety levels and compomer restoration color preferences was evaluated in 275 patients aged between 5 and 10 years who required restorative treatment in primary molar teeth. Children's dental anxiety levels were determined using the Modified Child Dental Anxiety Scale, face version (MCDAS-f). Children with identified anxiety levels were asked to choose colors for their fillings. A scale consisting of 9 colors (pink, blue, gold, silver, orange, yellow, green, purple, white) was used for color selection by adding white to the colored compomer scale.

ELIGIBILITY:
Inclusion Criteria:

* the child must be between 5-10 years old
* who needed restorative treatment of their deciduous molars
* no systemic disease or syndrome

Exclusion Criteria:

* the child is under 5 years old and over 10 years old
* who not needed restorative treatment of deciduous molars and haven't those teeth
* having any systemic disease or syndrome

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 275 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
anxiety level | before dental treatment to 30 minutes
  To determine the child's anxiety, the Modified Child Dental Anxiety Scale-faces version(MCDAS f) was administered to the children before restorative treatment. According to the MCDASf, a score was obtained by summing the scores of each question expressed with faces ranging from 1 "relaxed", 2 "slightly anxious", 3 "anxious", 4 "very anxious" and 5 "extremely anxious" according to 8 questions. A total score of less than 19 points was categorised as low anxiety, 19-31 points as moderate anxiety and 32-40 points as high anxiety.
colour preference | before dental treatment to 30 minutes
  The children were asked to choose from a new scale consisting of 9 colours (pink, blue, gold, silver, orange, yellow, green, purple, white) by adding white compomer (Dyract XP) to the colored compomer colour scale (Voco Twinky Star) for the compomer restoration color selections. During the color selection of the patients, it was ensured that the patients saw all the colors at the same time in order not to cause any guidance.
favorite color | before dental treatment to 30 minutes
  The patients were asked what their favourite color was after the compomer restoration color selection so that the previous question would not have any effect on the child's restoration color selection and the data obtained were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Edanur 1 çakır, Principal Investigator — Bülent Ecevit University
Locations (1):
- Bülent Ecevit Univercity, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No